CLINICAL TRIAL: NCT01910376
Title: Cancer in Elderly Nursing Home Residents in Belgium: Prospective Cohort Study Including Translational Research to Develop Better Prognostic Tools to Help With Treatment Decisions in the Elderly
Brief Title: Cancer in Nursing Home Residents
Status: Completed | Type: Observational
Sponsor: European Organisation for Research and Treatment of Cancer - EORTC (Network)
Collaborators: Armonea (Unknown)
Responsible Party: Sponsor
Other Study IDs: EORTC-1221
Record Dates: First submitted 2013-07-24; First posted 2013-07-29 (Estimated); Last update posted 2019-03-13 (Actual); Status verified 2019-03

CONDITIONS: Armonea Nursing Homes Residents

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Biospecimen Retention: Samples With DNA — Blood samples
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (3):
- Control cohort: Nursing home residents without cancer
- Cancer patient cohort: Patients in nursing homes with suspected or diagnosed active invasive cancer where a diagnostic or treatment decision has to be taken
- Biomarker cohort: Subgroup of individuals in the control cohort willing to provide a blood sample

SUMMARY:
Cancer is a disease of the elderly. Cancer incidence is 11-fold higher in persons over the age of 65, than in younger ones. Approximately 60% of all cancers and 70% of cancer mortality occurs in people older than 65 years. Moreover, due to the aging of the population in the Western world the number of elderly people is expected to increase and therefore the number of older cancer patients is expected to rise. Despite this rapid increase in cancer incidence and cancer-related mortality with age, our knowledge about ageing and cancer and about optimal treatment for older cancer patients is still far from adequate. Therefore, it is clear that cancer in the elderly is a major and increasing health problem. A key problem in geriatric oncology research is the important selection bias because very old/frail patients, are very rarely included in clinical trials.

Changes in the patterns of health care delivery have shifted the care of the elderly from acute care settings to the community and long-term care facilities. As the European population ages, more and more people will become nursing home residents, many of whom will have a suspicion of, or be diagnosed with, and eventually die from, cancer. Although cancer is very common in elderly nursing home residents, it is poorly studied. This lack of information may impact on clinical decision making and the appropriateness of treatments offered and therefore collection of this information is needed.

This project has two main objectives. The first objective is to report on demographics, referral patterns and motives for non-referral, anti-cancer treatments and outcome of patients in nursing homes with suspected or diagnosed active invasive cancer where a diagnostic or treatment decision has to be taken. The second objective is to develop better prognostic tools (for survival) including biological markers of ageing to help treatment decisions in the elderly.

ELIGIBILITY:
Inclusion Criteria:

All individuals:

* Age ≥ 65 years
* Residents in a nursing home in the Armonea network in Belgium.
* Absence of any psychological, familial, or sociological condition potentially hampering compliance with the study protocol; those conditions should be discussed with the patient/proxy before registration in the study.
* Written informed consent must be given according to ICH/GCP, and national/local regulations.
* The treating general practitioner (GP) is willing to provide medical information required by the study.

Cancer patient cohort:

Patients must have a new cancer event defined as one of:

* A strong clinical suspicion (based on physician's judgement) of a new cancer where a diagnostic or therapeutic decision needs to be taken.
* A strong clinical suspicion (based on physician's judgement) of progression of a previously known cancer where a diagnostic or therapeutic decision needs to be taken.
* Diagnosis of a new cancer where a diagnostic or therapeutic decision needs to be taken.
* Diagnosis of progression of a previously known cancer where a diagnostic or therapeutic decision needs to be taken.

All invasive cancer types and all histologies are eligible. All lines of treatment are eligible. Patients who are diagnosed with cancer during routine medical examinations for some other medical condition

Control cohort:

• Absence of known active invasive cancer, or strong clinical suspicion of cancer (based on physician's judgement) at baseline.

Exclusion criteria:

Patients who were not suspected to have cancer (progression) in the nursing home, but are hospitalized for other (medical) reasons, are then diagnosed with cancer during hospitalization.

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Study Population: Residents (≥ 65 years) in a nursing home in the Armonea network in Belgium.
Sampling Method: Non-Probability Sample
Enrollment: 125 (Actual)
Dates: Start 2014-10; Primary Completion 2017-12 (Actual); Study Completion 2017-12 (Actual)

PRIMARY OUTCOMES:
Prognostic capacity of p16INK4a expression in T lymphocytes on Overall Survival | The analyses will be performed when 90 deaths will have been observed
Demographics, referral patterns and motives for non-referral, anti-cancer treatments and outcome in nursing home patients with cancer or with strong clinical suspicion of cancer. | Baseline, every 3 months and for max. 2 years

SECONDARY OUTCOMES:
Comparison of baseline parameters and outcome between nursing home cancer patients (cancer patient cohort) and nursing home non-cancer patients (control cohort) | Baseline, every 3 months and for max. 2 years
Prognostic capacity of baseline clinical markers and Porock scale on OS, functional decline, cognitive decline and Quality of Life separately in nursing home cancer group (cancer patient cohort) and non-cancer group (control cohort). | Baseline, every 3 months and for max. 2 years
Prognostic capacity of other biomarkers of ageing on OS in the control group of nursing home patients without cancer. | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Hans Wildiers, Study Chair — UZ Leuven, Belgium
Locations (1):
- Armonea nursing homes network, Mechelen, Belgium